CLINICAL TRIAL: NCT00626132
Title: Evaluation of the Safety and Efficacy of a Standardized Eucommia Extract in the Treatment of Hypertension
Brief Title: Standardized Eucommia Extract in the Treatment of Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 25036
Record Dates: First submitted 2008-02-19; First posted 2008-02-29 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: Blood pressure; Herbs; Food
MeSH Terms: conditions — Hypertension | interventions — EAFP2 peptide, Eucommia ulmoides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eucommia (Experimental): Eucommia capsules two orally three times a day for 2 weeks
  Interventions: Dietary Supplement: Eucommia
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Eucommia

INTERVENTIONS:
Dietary Supplement: Eucommia — two capsules three times a day orally for 2 weeks

SUMMARY:
The purpose of this study is to demonstrate that eucommia, an herb used in China for making tea, is safe and effective for lowering blood pressure in humans with high blood pressure.

DETAILED DESCRIPTION:
Eucommia is an herb used as a tea in China and by traditional Chinese doctors to treat high blood pressure. People with high blood pressure in Russia were given eucommia with a reduction in blood pressure and without side effects. LSU Board of Regents supported this research to develop an herbal product that will maintain a healthy blood pressure. Dr. Liu with the LSU Ag Center extracted and standardized the eucommia. Dr. Baker with the LSU Vet School conducted safety studies in rats finding that eucommia was without side effects at 7 times the doses to be used in this study and there was a reduction in blood pressure in the rats. Dr. Greenway demonstrated that eucommia extract is a beta-adrenergic blocker, a mechanism used in approved blood pressure medications like propanolol.

Thirty healthy subjects will participate in this study who are between 18 and 70 years of age with less than 2 cardiovascular risk factors, and an average blood pressure of 120-160/80-100 on 3 screening visits to the Pennington Center clinic each a week apart. This level of high blood pressure can be safely treated with diet and lifestyle change alone for a 6 to 12-month period.

During screening subjects will come to the Pennington Center clinic on 3 occasions and have a medical history, physical examination, blood tests, and electrocardiogram (heart tracing) on 1 of these 3 visits, and 24-hour blood pressure monitoring. Visits will last approximately 30 minutes to 1 hour. If the subject is of childbearing potential, a pregnancy test will be done. A small box will be given to subjects that will be attached to a blood pressure cuff to carry on an arm for 24 hours on one occasion. This device will automatically take blood pressure every half hour during the 24-hour period.

Qualifying subjects return to the Pennington Center clinic on 3 occasions and will be asked to take 2 capsules 3 times a day for 2 weeks. The capsules could contain 1 gram of eucommia extract or a placebo (inactive sugar pill). Subjects have a 50:50 chance of receiving the eucommia and the assignment to eucommia or placebo will be made by chance (like flipping a coin). On each visit subjects will return the pill bottle, be given new medication to last until the next visit, be asked about any side effects, and have blood pressure taken. They will also be questioned about any adverse events. If blood pressure exceeds 180/110 on these visits, the subjects will be withdrawn from the trial and referred to their physician. At the end of the study, the blood tests, electrocardiogram, 24-hour blood pressure monitor, and physical examination will be repeated. These visits will last approximately 30 minutes to 1 hour, with the exception of visit 4 which will last approximately 1½ hours. The entire study will last approximately 5 weeks.

The effectiveness of eucommia in reducing blood pressure will be assessed by comparing the blood pressure readings from clinic visits and the 24-hour blood pressure monitoring. The safety of eucommia will be assessed from the blood tests, side effects, urinalysis, electrocardiogram, and physical examination. Subjects will be paid $35 per non-screening visit and an extra $30 for completing the study for a total of $100. At the end of the study or at the time of early termination, subjects will be instructed in the diet and lifestyle changes recommended by the National Institutes of Health and referred to their physicians.

There have been no side effects reported from taking eucommia and there was no toxicity in rats given the equivalent of 7 times the dose to be used in this trial. Drawing blood from an arm vein can cause discomfort from the needle, bruising, and rarely fainting or infection. These risks will be minimized by trained technicians and sterile technique. The 24-hour blood pressure monitor may be annoying and interrupt sleep when it automatically takes blood pressure.

ELIGIBILITY:
Eligible criteria:

* Are a healthy male or female
* Are 18 to 70 years of age
* Have a BMI (a number calculated from your height and weight) less than 40
* Have an average blood pressure measure between 120-160/80-100

Ineligible criteria:

* Smoke or have smoked in the past 6 months
* Have diabetes mellitus
* Have heart disease including left ventricular hypertrophy, prior myocardial infarction (heart attack), angina pectoris (heart pain), a prior revascularization procedure (heart bypass), heart failure or stroke
* Have nephropathy (kidney disease)
* Have peripheral arterial disease (blockage of the arteries to your body)
* Have retinopathy (disease of the back of the eye)
* Take a beta-adrenergic blocking drug
* Regularly use medications that would influence weight, or unstable doses of medicines that would affect blood pressure
* Are pregnant or nursing a baby
* Are taking blood pressure medications and not on a stable dose for 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure and ambulatory monitor | After 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States